CLINICAL TRIAL: NCT00424190
Title: A Phase 3, Multicenter, Randomized, Double-blind, Comparative Study to Evaluate the Safety and Efficacy of Ceftaroline Versus Vancomycin Plus Aztreonam in Adult Subjects With Complicated Skin and Skin Structure Infection
Brief Title: Comparative Study of Ceftaroline vs. Vancomycin Plus Aztreonam in Adult Subjects With Complicated Skin Infections
Acronym: cSSSI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Senior Vice President, Clinical Development, Cerexa, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P903-06
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Results first posted 2010-11-08 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Bacterial Infections
Keywords: Abscess; Antibacterial; Antibiotic; Antimicrobial; Bacterial infection, skin; Ceftaroline; Ceftaroline acetate; Cellulitis; Cephalosporin; Complicated skin and skin structure infection; cSSSI; Intravenous; Methicillin-resistant Staphylococcus Aureus (MRSA); PPI-0903; Prodrug; Skin disease, bacterial; Skin infection; Staphylococcal skin infection; Staphylococcus aureus; Streptococcal skin infection; Surgical site infection; TAK-599
MeSH Terms: conditions — Bacterial Infections; Abscess; Skin Diseases, Bacterial; Cellulitis; Staphylococcal Skin Infections; Staphylococcal Infections; Surgical Wound Infection | interventions — Vancomycin; Aztreonam; Ceftaroline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ceftaroline for Injection (Experimental)
  Interventions: Drug: Ceftaroline
- IV Vancomycin and IV Aztreonam (Active Comparator)
  Interventions: Drug: IV Vancomycin plus IV Aztreonam

INTERVENTIONS:
Drug: IV Vancomycin plus IV Aztreonam — vancomycin at 1 g parenteral infused over 60 minutes followed by aztreonam 1 g infused over 60 minutes, every 12 hours, for 5 to 14 days.
  Other Names: Active Comparator
  Arms: IV Vancomycin and IV Aztreonam
Drug: Ceftaroline — 600 mg parenteral infused over 60 minutes, every 12 hours for 5 to 14 days
  Other Names: Experimental
  Arms: Ceftaroline for Injection

SUMMARY:
The purpose of this study is to determine whether ceftaroline is effective and safe in the treatment of complicated skin infections in adults.

DETAILED DESCRIPTION:
Additional purpose of the study is to compare ceftaroline effectivity versus Vancomycin plus Aztreonam in the treatment of complicated skin infections in adults.

ELIGIBILITY:
Inclusion Criteria:

* Skin and skin structure infection (SSSI) that involves deeper soft tissue or requires significant surgical intervention, or cellulitis or abscess on lower extremity which occurs in subjects with diabetes mellitus or well-documented peripheral vascular disease.

Exclusion Criteria:

* Prior treatment of current cSSSI with an antimicrobial.
* Failure of vancomycin or aztreonam as therapy for the current cSSSI, or prior isolation of an organism with in vitro resistance to vancomycin or aztreonam.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 698 (Actual)
Dates: Start 2007-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Corey, MD, Principal Investigator — Duke University
Locations (44):
- United States (14):
  - Investigational Site, Dothan, Alabama
  - Investigational Site, Long Beach, California
  - Investigational Site, Los Angeles, California
  - Investigational Site, Sacramento, California
  - Investigational Site, San Diego, California
  - Investigational Site, San Francisco, California
  - Investigational Site, Torrance, California
  - Investigational Site, Savannah, Georgia
  - Investigational Site, Naperville, Illinois
  - Investigational Site, Indianapolis, Indiana
  - Investigational Site, Shreveport, Louisiana
  - Investigational Site, Columbus, Ohio
  - Investigational Site, Landsdale, Pennsylvania
  - Investigational Site, Tacoma, Washington
- Argentina (6):
  - Investigational Site, Buenos Aires
  - Invetigational Site, Buenos Aires
  - Investigational Site, Córdoba
  - Invetigational Site, Córdoba
  - Investigational Site, Entre Ríos
  - Investigational Site, Santa Fe
- Brazil (2):
  - Investigational Site, Curiuba-Parans
  - Investigational Site, São Paulo
- Chile (2):
  - Investigational Site, Santiago
  - Investigational Site, Viña del Mar
- Germany (5):
  - Investigational Site, Berlin
  - Investigational Site, Bochum
  - Investigational Site, Hanau
  - Investigational Site, Plauen
  - Investigational Site, Quedlinburg
- Investigational Site, Chihuahua City, Mexico
- Invetigational Site, Lima, Peru
- Poland (5):
  - Investigational Site, Bytom
  - Investigational Site, Krakow
  - Investigational Site, Lublin
  - Investigational Site, Sosnowiec
  - Investigational Site, Todz
- Romania (2):
  - Investigational Site, Bucharest
  - Investigational Site, Timișoara
- Russia (3):
  - Investigational Site, Moscow
  - Investigational Site, Saint Petersburg
  - Investigational Site, Smolensk
- Ukraine (3):
  - Investigational Site, Dnipropetrovsk
  - Investigational Site, Ivano-Frankivsk
  - Investigational Site, Lviv

REFERENCES:
- [Derived] Dryden M, Kantecki M, Yan JL, Stone GG, Leister-Tebbe H, Wilcox M. Treatment outcomes of secondary bacteraemia in patients treated with ceftaroline fosamil: pooled results from six phase III clinical trials. J Glob Antimicrob Resist. 2022 Mar;28:108-114. doi: 10.1016/j.jgar.2021.10.027. Epub 2021 Dec 16. PMID 34922058
- [Derived] Wilcox M, Yan JL, Gonzalez PL, Dryden M, Stone GG, Kantecki M. Impact of Underlying Comorbidities on Outcomes of Patients Treated with Ceftaroline Fosamil for Complicated Skin and Soft Tissue Infections: Pooled Results from Three Phase III Randomized Clinical Trials. Infect Dis Ther. 2022 Feb;11(1):217-230. doi: 10.1007/s40121-021-00557-w. Epub 2021 Nov 6. PMID 34741280
- [Derived] Corey GR, Wilcox MH, Gonzalez J, Jandourek A, Wilson DJ, Friedland HD, Das S, Iaconis J, Dryden M. Ceftaroline fosamil therapy in patients with acute bacterial skin and skin-structure infections with systemic inflammatory signs: A retrospective dose comparison across three pivotal trials. Int J Antimicrob Agents. 2019 Jun;53(6):830-837. doi: 10.1016/j.ijantimicag.2019.01.016. Epub 2019 Feb 1. PMID 30716446
- [Derived] Cheng K, Pypstra R, Yan JL, Hammond J. Summary of the safety and tolerability of two treatment regimens of ceftaroline fosamil: 600 mg every 8 h versus 600 mg every 12 h. J Antimicrob Chemother. 2019 Apr 1;74(4):1086-1091. doi: 10.1093/jac/dky519. PMID 30597021
- [Derived] Corrado ML. Integrated safety summary of CANVAS 1 and 2 trials: Phase III, randomized, double-blind studies evaluating ceftaroline fosamil for the treatment of patients with complicated skin and skin structure infections. J Antimicrob Chemother. 2010 Nov;65 Suppl 4:iv67-iv71. doi: 10.1093/jac/dkq256. PMID 21115456
- [Derived] Corey GR, Wilcox MH, Talbot GH, Thye D, Friedland D, Baculik T; CANVAS 1 investigators. CANVAS 1: the first Phase III, randomized, double-blind study evaluating ceftaroline fosamil for the treatment of patients with complicated skin and skin structure infections. J Antimicrob Chemother. 2010 Nov;65 Suppl 4:iv41-51. doi: 10.1093/jac/dkq254. PMID 21115454
- [Derived] Corey GR, Wilcox M, Talbot GH, Friedland HD, Baculik T, Witherell GW, Critchley I, Das AF, Thye D. Integrated analysis of CANVAS 1 and 2: phase 3, multicenter, randomized, double-blind studies to evaluate the safety and efficacy of ceftaroline versus vancomycin plus aztreonam in complicated skin and skin-structure infection. Clin Infect Dis. 2010 Sep 15;51(6):641-50. doi: 10.1086/655827. PMID 20695801

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited worldwide from February 2007 to November 2007
Pre-assignment Details: Patients were screened for up to 24 hours
Groups:
- Ceftaroline Fosamil for Injection: Ceftaroline fosamil 600 mg administered IV over 60 minutes every 12 hours followed by placebo administered over 60 minutes every 12 hours
- IV Vancomycin Plus IV Aztreonam: Vancomycin 1 g administered over 60 minutes every 12 hours followed by aztreonam 1 g administered over 60 minutes every 12 hours
Period: Overall Study
Arm/Group | Ceftaroline Fosamil for Injection | IV Vancomycin Plus IV Aztreonam
Started | 351 | 347
Completed | 329 | 317
Not Completed | 22 | 30
Not completed — Withdrew consent | 3 | 4
Not completed — Death | 3 | 0
Not completed — Noncompliance | 1 | 2
Not completed — Request of sponsor or investigator | 0 | 2
Not completed — Diagnosis of osteomyelitis | 0 | 1
Not completed — Other | 15 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftaroline Fosamil for Injection | IV Vancomycin Plus IV Aztreonam | Total
Number analyzed (Participants) | 351 | 347 | 698
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (17.17) | 47.2 (17.01) | 48.2 (17.10)
Age, Customized [Number; unit: participants]
  >=65 years | 57 | 72 | 129
  <18 years | 0 | 0 | 0
  >=18 years and < 65 years | 294 | 275 | 569
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 129 | 260
  Male | 220 | 218 | 438
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic | 268 | 270 | 538
  Hispanic | 83 | 77 | 160

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure Rate at Test of Cure (TOC) (MITT Population)
Description: Cure: Total resolution of all signs and symptoms of the baseline infection, or improvement of the infection such that no further antimicrobial therapy was necessary.
  Failure: Requirement of alternative antimicrobial therapy for primary infection of cSSSI due to inadequate response, recurrence, new infection at the same site; treatment-limiting adverse event (AE); requirement for surgery due to failure of study drug; diagnosis of osteomyelitis after Study Day 8; or death caused by cSSSI.
  Indeterminate: Inability to determine an outcome
Time Frame: 8-15 days after the end of treatment
Population: MITT (Modified Intent to Treat) - Any randomized subjects that received any amount of study drug
Measure: Number; unit: participants
Arm/Group | Ceftaroline Fosamil for Injection | IV Vancomycin Plus IV Aztreonam
Number analyzed (Participants) | 351 | 347
participants
  Clinical Cure | 304 | 297
  Clinical Failure | 29 | 21
  Indeterminate | 18 | 29
Statistical Analysis 1: Comparison: Ceftaroline Fosamil for Injection vs IV Vancomycin Plus IV Aztreonam; The primary objective of this study was to determine the noninferiority in clinical cure rate of ceftaroline in comparison with vancomycin plus aztreonam in adult subjects with cSSSI; Test type: Non-Inferiority or Equivalence — A two-sided 95% confidence interval (CI) for the observed difference in the primary outcome measure between ceftaroline and vancomycin plus aztreonam was calculated. Noninferiority was concluded if the lower limit of the 95% CI was higher than -10%; Risk Difference (RD) = 1.0, 95% CI 2-sided [-4.2 to 6.2] — Risk difference corresponds to Ceftaroline clinical cure rate minus Vancomycin plus Aztreonam clinical cure rate. The confidence interval was calculated using the Miettinen and Nurminen method without adjustment

2. Primary Outcome: Clinical Cure Rate of Ceftaroline Compared With That of Vancomycin Plus Aztreonam Treatment at TOC in the Clinically Evaluable (CE) Population
Time Frame: 8-15 days after last dose of study drug
Reporting Status: Not Posted

3. Secondary Outcome: Microbiological Success Rate at the TOC Visit
Time Frame: 8-15 days after last dose of study drug
Reporting Status: Not Posted

4. Secondary Outcome: Clinical Response at the End of Therapy (EOT) Visit
Time Frame: Last day of study drug administration
Reporting Status: Not Posted

5. Secondary Outcome: Clinical and Microbiological Response by Pathogen at the TOC Visit
Time Frame: 8-15 days after last dose of study drug
Reporting Status: Not Posted

6. Secondary Outcome: Clinical Relapse at the Late Follow Up (LFU) Visit
Time Frame: 21 to 35 days after the last dose of study drug
Reporting Status: Not Posted

7. Secondary Outcome: Microbiological Reinfection or Recurrence at the LFU Visit
Time Frame: 21 to 35 days after the last dose of study drug
Reporting Status: Not Posted

8. Secondary Outcome: Assess Safety
Description: Comparisons of the number of participants with Adverse Events
Time Frame: First dose of study drug through TOC visit
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: All safety analysis was performed on the Safety Population, those subjects that had received any amount of the actual study drug.
Arm/Group | Ceftaroline Fosamil for Injection | IV Vancomycin Plus IV Aztreonam
Serious Adverse Events (participants affected / at risk) | 16/351 | 12/347
Other Adverse Events (participants affected / at risk) | 128/351 | 162/347
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftaroline Fosamil for Injection (N=351) | IV Vancomycin Plus IV Aztreonam (N=347)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Generalized edema (General disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Electrocardiogram ST segment elevation (Investigations) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arterial thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftaroline Fosamil for Injection (N=351) | IV Vancomycin Plus IV Aztreonam (N=347)
Nausea (Gastrointestinal disorders) | 20 (20) | 16 (16)
Headache (Nervous system disorders) | 18 (18) | 13 (13)
Pruritus generalized (Skin and subcutaneous tissue disorders) | 13 (13) | 16 (16)
Diarrhea (Gastrointestinal disorders) | 12 (12) | 11 (11)
Rash (Skin and subcutaneous tissue disorders) | 12 (12) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (11) | 29 (29)
Vomiting (Gastrointestinal disorders) | 9 (9) | 9 (9)
Constipation (Gastrointestinal disorders) | 8 (8) | 6 (6)
Dizziness (Nervous system disorders) | 8 (8) | 6 (6)
Insomnia (Psychiatric disorders) | 5 (5) | 9 (9)
Pyrexia (General disorders) | 4 (4) | 9 (9)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 9 (9)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 7 (7)
Fatigue (General disorders) | 1 (1) | 7 (7)
Hypertension (Vascular disorders) | 1 (1) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No